CLINICAL TRIAL: NCT06808958
Title: The Effect of Bathtub Bath on Stress and Comfort in Infants Receiving Phototherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Necla Kasımoğlu, Assistant Professor, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 124567
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Bathtub Bath
Keywords: Bathtub Bath; Infants; Phototherapy
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The newborn's eyes will be covered with a phototherapy eye patch and placed in the baby's jeans and the treatment will be started. The position (face down and back down) is changed every two hours. And phototherapy is paused every three hours for feeding. Therefore, the bath will be given half an hour after the phototherapy application is completed before the two phototherapy sessions. The physiological parameters of the newborns will be evaluated 0 minutes before the bath. Then the bathtub bath application will be started. The bath application will be completed in a time not exceeding 5 minutes. Physiological parameters, stress and comfort will be assessed 15 minutes after bathing. Then, 15 minutes after starting the phototherapy session and 15 minutes before ending the phototherapy session, physiological parameters, stress and comfort will be assessed. The measured physiological parameters (respiratory rate, heart rate, oxygen saturation and body temperature), stress and comfort scor
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Bathtub Bath) Group (Experimental): The newborn's eyes will be covered with a phototherapy eye patch and placed in the baby's jeans and the treatment will be started. Therefore, the bath will be given half an hour after the phototherapy application is completed before the two phototherapy sessions. The physiological parameters of the newborns will be evaluated 0 minutes before the bath. Then the bathtub bath application will be started. The bath application will be completed in a time not exceeding 5 minutes. Physiological parameters, stress and comfort will be assessed 15 minutes after bathing. Then, 15 minutes after starting the phototherapy session and 15 minutes before ending the phototherapy session, physiological parameters, stress and comfort will be assessed. The measured physiological parameters (respiratory rate, heart rate, oxygen saturation and body temperature), stress and comfort stress and comfort scores will be recorded on the Newborn Follow-up Form.
  Interventions: Behavioral: Experimental (Bathtub Bath) Group
- Control Group (No Intervention): nformation about the newborns selected for the control group (gender of the baby, gestational week, delivery method, etc.) will be taken from the newborn file and recorded on the form containing the newborn's introductory information. Physiological parameter, stress and comfort assessments will be performed on the newborns in the control group without any different application, immediately before the phototherapy session starts, 0 minutes before, 15 minutes after starting and 15 minutes before the phototherapy session ends. The measured physiological parameters (respiratory rate, heart rate, oxygen saturation and body temperature), stress and comfort scores will be recorded on the Newborn Follow-up Form.

INTERVENTIONS:
Behavioral: Experimental (Bathtub Bath) Group — The newborn's eyes will be covered with a phototherapy eye patch and placed in the baby's jeans and the treatment will be started. The position (face down and back down) is changed every two hours. And phototherapy is paused every three hours for feeding. Therefore, the bath will be given half an hour after the phototherapy application is completed before the two phototherapy sessions. The physiological parameters of the newborns will be evaluated 0 minutes before the bath. Then the bathtub bath application will be started. The bath application will be completed in a time not exceeding 5 minutes. Physiological parameters, stress and comfort will be assessed 15 minutes after bathing. Then, 15 minutes after starting the phototherapy session and 15 minutes before ending the phototherapy session, physiological parameters, stress and comfort will be assessed. The measured physiological parameters (respiratory rate, heart rate, oxygen saturation and body temperature), stress and comfort scor
  Arms: Experimental (Bathtub Bath) Group

SUMMARY:
After intrauterine life, intensive care is a stressful environment for newborns who have to start their lives in the NICU. Many care practices in the NICU, including environmental factors (such as light, sound), heel prick blood collection, routine care, invasive interventions and bathing, are sources of stress for newborns. At the same time, the physical structure of the NICU, that is, factors such as sound, light, odor, and the physiological and anatomical immaturity of newborn babies, routine care and invasive procedures can reduce the comfort of the baby. Controlling the factors that may cause stress in the infant in the NICU and reducing stress and increasing comfort at the same time may affect the baby's healing process and discharge process.

Recently, nursing care practices that reduce stress and increase comfort are at the forefront and have become an important concept today. In the literature, massage, kangaroo care, swaddling, listening to the mother's voice, listening to music, positioning, mother-scented hand simulation, breastfeeding, wrapping, bathing . Neonatal bathing is among the practices frequently performed by neonatal intensive care nurses to reduce the stress of the newborn and increase comfort Bathing is a basic skin care process for newborns. Bathing is known to have beneficial effects for infants. It is reported that bathing causes relaxation in muscles, is calming and relaxing, is effective in regulating body temperature and reducing pain, regulating blood circulation and respiratory system, and supporting parent-infant bonding (interaction).

Bathing is a basic skin care process for newborns. Bathing is known to have beneficial effects for infants. It is reported that bathing causes relaxation in muscles, is calming and relaxing, is effective in regulating body temperature and reducing pain, regulating blood circulation and respiratory system, and supporting parent-infant bonding (interaction). Bowles (2013) found that neonatal bathing exfoliates dead skin cells, re-moisturizes the skin surface, reduces infant stress and agitation to provide comfort, encourages flexion and containment, and eventually provides developmentally supportive care. In the literature, there are many studies showing that bathing is also effective in reducing bilirubin levels in infants hospitalized with hyperbilirubinemia in neonatal intensive care units.

Stimuli such as lighting, noise and pain from repeated medical interventions in the NICU can cause stress in infants. Excessive lighting can cause negative effects such as weight gain disorder, sleep disturbance and stress in infants. Since phototherapy light is not only a source of stress for the baby receiving phototherapy but also one of the important factors affecting the comfort level, the comfort of babies receiving phototherapy should be monitored frequently. The physical conditions of NICUs, physiologic and anatomic conditions of the infants receiving treatment, invasive interventions and care lead to a decrease in the comfort level of newborns. This situation negatively affects the discharge time and recovery of newborns. Therefore, this study will be conducted to examine the effect of bathtub bathing on stress level and comfort in infants receiving phototherapy in neonatal intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with a gestational age of 37 weeks and above
* Birth weight of 2500 grams and above
* Having completed 24 hours after birth
* The newborn is hospitalized with a diagnosis of physiological hyperbilirubinemia and is receiving phototherapy
* No accompanying disease
* No accompanying treatment
* Stable physiological parameters (no tachycardia and bradycardia)
* No respiratory failure or distress (respiratory rate between 30-60, not being monitored on a ventilator, oxygen saturation of 90% and above, no need for continuous high concentration oxygen with methods such as Hood, CPAP, etc.)
* The baby is hospitalized during data collection
* The parents are willing for the newborn to participate in the study Exclusion Criteria
* Preterms with a gestational age of 22-37 weeks,
* The newborn has another concomitant disease diagnosis
* Has been wiped or bathed in a tub within the last 12 hours
* Has been hospitalized with a diagnosis of pathological hyperbilirubinemia
* Has been given sedatives and/or muscle relaxants
* The parent does not want the newborn to participate in the study or wants/wants to withdraw from the study while the study is ongoing

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Newborn Stress Scale | Physiological parameters, stress and comfort will be assessed 15 minutes after bathing. Then, 15 minutes after starting the phototherapy session and 15 minutes before ending the phototherapy session, 0 minutes before, 15 minutes after starting and 15 min
  The Newborn Stress Scale (NSS), developed by Ceylan and Bolışık (2017), consists of a total of 24 items on a 3-point Likert scale. The scale items include 8 subgroups including facial expression, body color, respiration, activity level, comfortability, muscle tone, extremities, and posture, and each subgroup is evaluated between 0-2 points in the scoring. The minimum score is zero and the maximum score is 16 points. As the score increases, the baby's stress level increases.

SECONDARY OUTCOMES:
Newborn Comfort Behavior Scale | 0 minutes before, 15 minutes after starting and 15 minutes before the phototherapy session ends. stress and comfort will be assessed 15 minutes after bathing. Then, 15 minutes after starting the phototherapy session and 15 minutes before ending the photo
  The scale is a Likert-type scale developed to be used in the evaluation of sedation and comfort needs, pain and distress of newborns monitored in intensive care. Van Dijk et al. In 2009, the scale was revised and the COMFORTneo scale was validated and its reliability was established to measure only behavior in newborns without physiological parameters. The Neonatal Comfort Behavior Scale (NCBSS), whose validity and reliability were established by Kahraman, Başbakkal and Yalaz (2014), is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension and muscle tone.

IPD SHARING:
Plan to Share IPD: No